### CLINICAL STUDY PROTOCOL



# Protocol Title: A Phase 3, Multicenter, Randomized, Double-Blind, Placebo-Controlled Study to Assess the Efficacy and Safety of REL-1017 for Treatment of Major Depressive Disorder (The RELIANCE-I Study)

Protocol Number: REL-1017-301

NCT Number: NCT04688164

Name of Investigational Product: REL-1017

Phase of Development: 3

Indication: Major Depressive Disorder Sponsor: Relmada Therapeutics Inc.

Document Date: December 01 2022

Certain information within this protocol has been redacted to protect either personally identifiable information or company confidential information.

This may include, but is not limited to, redaction of the following:

- Names, addresses, and other personally identifiable information
- Proprietary information, such as scales or coding systems, which are considered confidential information.
- Other information as needed to protect the trade secret and/or confidential information of Relmada Therapeutics

### CLINICAL STUDY PROTOCOL



# Protocol Title: A Phase 3, Multicenter, Randomized, Double-Blind, Placebo-Controlled Study to Assess the Efficacy and Safety of REL-1017 for Treatment of Major Depressive Disorder (The RELIANCE-I Study)

Protocol Number: REL-1017-301

| Name of Investigational Product: | REL-1017 |
|---|---|
| Phase of Development: | 3 |
| Indication: | |
| Sponsor: | Relmada Therapeutics, Inc. 2222 Ponce de Leon Blvd, Floor 3 |
| | Coral Gables, FL 33134 |
| Protocol Version: | |
| Amendment Version: | |
| Protocol Date: | December 01 2022 |

### -CONFIDENTIAL-

This document and its contents are the property of and confidential to Relmada Therapeutics, Inc. Any unauthorized copying or use of this document is prohibited.

### PROTOCOL APPROVAL SIGNATURES

| III O I O O O D I III I II O | , 122 5151 121 5125 |
|---|---|
| Protocol Title: | A Phase 3, Multicenter, Randomized, Double-Blind, Placebo-<br>Controlled Study to Assess the Efficacy and Safety of REL-1017 for<br>Treatment of Major Depressive Disorder (The RELIANCE-I Study) |
| Protocol Number: | REL-1017-301 |
| Protocol Version | |
| Amendment Version | |
| This study will be conducted in compliance with the clinical study protocol (and amendments), International Council for Harmonisation (ICH) guidelines for current Good Clinical Practice (GCP), and applicable regulatory requirements. Sponsor Signatory Signature Signature Date (DD-Mmm-YYYY) | |

### INVESTIGATOR SIGNATURE PAGE

**Protocol Title:** A Phase 3, Multicenter, Randomized, Double-Blind, Placebo-Controlled

Study to Assess the Efficacy and Safety of REL-1017 for Treatment of

Major Depressive Disorder (The RELIANCE-I Study)

**Protocol Number:** REL-1017-301

## Confidentiality and Current Good Clinical Practice (GCP)/E6(R2):

I agree, as an Investigator conducting this study:





## 1 SYNOPSIS

| Title of Study | Study to Assess | icenter, Randomized, Double-Blind, Placebo-Controlled<br>the Efficacy and Safety of REL-1017 for Treatment of<br>re Disorder (The RELIANCE-I Study) |
|---|---|---|
| Sponsor | Relmada Therapeutics, Inc. (Relmada) | |
| Investigators/Study Sites | Approximately | planned in the United States |
| Phase of Development | 3 | |

| Objectives | Endpoints |
|---|---|
| Primary | |
| To evaluate the therapeutic efficacy of REL-<br>1017 in subjects with inadequate response to<br>ongoing antidepressant therapy (ADT)compared<br>to placebo at Day 28 on the Montgomery-<br>Åsberg Depression Rating Scale (MADRS10)<br>total score<br><b>Key Secondary</b> | Absolute change from Baseline to Day 28 of the MADRS10 total score in REL-1017 compared to placebo in subjects with inadequate response to ongoing ADT |
| <ul> <li>Key Secondary Efficacy Objectives</li> <li>To evaluate the therapeutic efficacy of REL-1017 for treatment of Major Depressive Disorder (MDD) in subjects with inadequate response to ongoing ADT compared to placebo in the following measurements: <ul> <li>Clinical Global Impression of Severity (CGI-S) score at Day 28</li> <li>MADRS10 score at Day 7</li> <li>MADRS10 remission rate (total score ≤10) at Day 28</li> <li>MADRS10 response rate (improvement ≥50% compared with total Baseline score) at Day 28</li> </ul> </li> </ul> | <ul> <li>CGI-S score</li> <li>Absolute change from Baseline to Day 7 of the MADRS10 total score</li> <li>MADRS10 remission rate (total score ≤10) at Day 28</li> <li>MADRS10 response rate (improvement ≥50% compared with total Baseline score) at Day 28</li> </ul> |



| Objectives | Endpoints |
|---|---|
| Safety | |
| Safety and Tolerability Objectives To evaluate safety and tolerability of REL-1017 | <ul> <li>Treatment-emergent adverse events (TEAEs)</li> <li>Vital signs and weight</li> <li>Physical examination</li> <li>Clinical laboratory parameters (chemistry, hematology, and urinalysis)</li> <li>C-SSRS</li> </ul> |
| Pharmacokinetic | |
| Pharmacokinetic Objectives • To evaluate pharmacokinetics (PK) of REL-1017 and potential metabolites | Estimation of REL-1017 PK profile (maximum observed plasma concentration [C <sub>max</sub> ], trough concentration [C <sub>trough</sub> ], and apparent terminal elimination half-life at steady state [t <sub>1/2</sub> ] based on sparse PK sampling |

| Study Design | This is an outpatient, 2-arm, Phase 3, multicenter, randomized, double-blind, placebo-controlled study to assess the efficacy and safety of REL-1017 at 25 mg once daily (QD) for treatment of MDD in subjects with inadequate response to ongoing ADT |
|---|---|
| Investigational<br>Product/Reference Product | REL-1017 in 25 mg and matching placebo |
| Study Drug, Dose Schedule,<br>and Mode of<br>Administration | REL-1017 in a 25 mg tablet for oral administration by mouth (PO) The following dose schedule will be used in the study: |
| | Day 1 – loading dose: Three REL-1017 25 mg tablets (75 mg total) administered at the clinical study site Three matching placebo tablets administered at the clinical study site |
| | Day 2 to Day 28 – maintenance dose: One REL-1017 25 mg tablet QD One matching placebo tablet QD |

Participants will be asked to stay on a stable dosing regimen of the current antidepressant therapy (ADT) between Day 1 and Day 28, while exposed to REL-1017 or matching placebo. Dosing with REL-1017 should take place once daily at the same time as the first-line ADT is taken. Adult participants (aged 18 to 65 years, inclusive) diagnosed with MDD Study Population and (based on Structured Clinical Interview for DSM-5 [SCID-5] for MDD, **Duration of Participation** matching Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition [DSM-5]), who are currently in a major depressive episode (MDE), and with a substantiated inadequate response to 1 to 3 courses of a valid course of an approved antidepressant in the current MDE, ie, to an approved dose and duration (minimum 6 weeks) of a marketed ADT treatment course The maximum duration of the MDE must not exceed 36 months. After signing of the informed consent form (ICF), each participant will undergo an up to 30-day Screening period and a 28-day randomized double-blind placebo-controlled period, for a total of approximately 58 days of study participation. For approximately the first 200 completers of the 28-day dosing with study drug, a 14-day safety follow-up period will be added, extending the time of study participation to approximately 72 days. All participants who complete the 28-day treatment period will be offered the opportunity to enroll in a 1 year open-label study under its separate study protocol. Planned Sample Size The REL-1017-301 study is designed to achieve 90% power, with an overall two-tailed  $\alpha$ -level of 0.05.



#### **Inclusion Criteria**

To enroll in the clinical study, participants must meet the following inclusion criteria:

- Must be able to read, speak, and understand English or Spanish and must provide written informed consent prior to the initiation of any protocol-specific procedures.
- 2. Male or female participant, aged 18 to 65 years, inclusive.

3.

- Participant is willing and able to commit to meet all study requirements, adhere to both approved ADT and study drug regimen, and complete all assessments and all scheduled visits, per Investigator judgment.
- 5. Women of childbearing potential (WOCBP) and men whose sexual partners are WOCBP must use at least 1 highly effective method of contraception from Screening and for at least 2 months after the last study drug administration. For men with female sexual partners of childbearing potential, examples of medically acceptable forms of contraception include vasectomy or male condom for participants, plus an additional method of contraception for their female partners. Highly effective methods of contraception are those which have a failure rate of <1% (when implemented consistently and correctly) and include:
  - Intrauterine device (IUD)
  - Bilateral tubal ligation, bilateral salpingectomy, or bilateral tubal occlusive procedure
  - Hormonal contraceptives (eg, oral, patch, or injectable)
  - A double-barrier protection method (eg, condom, sponge, or vaginal diaphragm with spermicide cream, foam, or gel)
  - Abstinence from heterosexual intercourse is accepted if this is the participant's usual lifestyle and must be continued until at least 2 months after the last dose of study drug.

Women who are not of childbearing potential must be congenitally or surgically sterile (hysterectomy and/or bilateral

- oophorectomy/salpingo-oophorectomy, as determined by the participant's medical history) or must be post-menopausal. Post-menopausal is defined as being amenorrheic for at least 1 year without another cause and a follicle-stimulating hormone (FSH) level ≥40 mIU/mL as confirmation.
- 6. Diagnosed with MDD as defined by the Diagnostic and Statistical Manual, Fifth Edition (DSM-5), and confirmed by the SCID-5 MDD.
- 7. Hamilton Depression Rating Scale-17 (HAMD17) score at Screening and independently confirmed by SAFER assessment.
- Diagnosed with a current MDE lasting from 8 weeks to 36 months as
  defined by the DSM-5 and confirmed by the SCID-5 MDD, as well as
  independent confirmation of HAMD17 score, SAFER/ATRQ, and
  contextual appropriateness to be a participant in this study, after
  evaluation by an MGH-CTNI clinician.
- 10. Treated for at least 6 weeks prior to Screening and stabilized for at least 6 weeks prior to Baseline on an approved dosing regimen of ADT (eg, selective serotonin reuptake inhibitor [SSRI], serotonin and norepinephrine reuptake inhibitor [SNRI], bupropion (a norepinephrine–dopamine reuptake inhibitor [NDRI] and nicotinic receptor antagonist) during the current MDE, and committed to remaining on the same stable dosing regimen for the Screening period and for the entire study, at or above the minimally adequate dose in the ATRQ. Maximal doses and recommended doses for each ADT are at the discretion of the Investigator and Medical Monitor, except for citalopram and escitalopram

**Exclusion Criteria** 

 History or presence of clinically significant abnormality as assessed by physical examination, medical history, 12-lead ECG, vital signs, or laboratory values, which in the opinion of the Investigator would jeopardize the safety of the participant or the validity of the study

- results, including established QT prolongation, long QT syndrome, torsades de pointes, bradyarrhythmia, ventricular tachycardia, uncompensated heart failure (greater than New York Heart Association [NYHA] Class 1 congestive heart failure [CHF]), uncontrolled hypokalemia, or uncontrolled hypomagnesemia.
- 2. More than class 2 angina pectoris or a myocardial infarction (MI) or acute coronary syndrome within the past 3 months.
- Any medical, psychiatric condition, or social context that, in the
  opinion of the investigator, is likely to unfavorably alter the riskbenefit of subject participation, to interfere with protocol compliance,
  or to confound safety or efficacy assessments.
- 4. Have any significant illness, of any nature, including possible Coronavirus-SARS-2 related fever and symptoms, requiring hospitalization, emergency treatment, or isolation (quarantine) within 4 weeks prior to Screening or during the Screening period, and as determined by the Investigator.
- 5. History or first degree relative with history of unexplained sudden death or long QT syndrome.
- Triplicate 12-lead ECG with average QTcF (QT interval with Fridericia's correction) ≥450 msec and/or a QRS interval ≥120 msec at Screening.
- 7. Current or recent uncontrolled orthostasis or orthostatic hypotension necessitating treatment.
- 8. Poorly controlled diabetes as defined by a glycosylated hemoglobin (HbA1c) >7.5%, despite standard care.
- Any use of long-term prescribed opioids (ie, >120 days in a 6-month period) within 6 months prior to Screening or any recreational use of opioids.
- 12. Use of any anxiolytic, antipsychotic, anticonvulsant/antiepileptic, mood stabilizer, or stimulant medication(s) within 30 days prior to Baseline. Note: Participant should be medically stable, the medication was appropriately tapered and participant has no withdrawal symptoms.
- 13. Use of St. John's Wort, [Hypericum Perforatum]) within 30 days prior to Baseline.
- 14. Participated in a ketamine, esketamine, dextromethorphan or any other NMDAR-antagonist study, or who received esketamine at any time.
- 15. Received ketamine, memantine, and/or dextromethorphan treatment within 30 days prior to Screening.
- 16. History of allergy or hypersensitivity to methadone or related drugs.
- Receiving new-onset psychotherapy (individual, group, marriage, or family therapy) within 2 months prior to Screening, or planning to start psychotherapy at any time during participation in the study.
- Any lifetime experience of electroconvulsive therapy (ECT) and/or vagus nerve stimulation (VNS), or any other type of physical brain stimulation.
- 19. Received repetitive transcranial magnetic stimulation (rTMS) less than 6-months prior to the Screening visit.



